CLINICAL TRIAL: NCT04605926
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Itolizumab in Subjects Hospitalized With COVID-19
Brief Title: A Study to Evaluate the Efficacy and Safety of Itolizumab in Subjects Hospitalized With COVID-19
Acronym: EQUINOX
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor has currently elected to withhold study initiation
Sponsor: Equillium (Industry)
Collaborators: Biocon Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EQ001-20-001
Record Dates: First submitted 2020-10-21; First posted 2020-10-28 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Coronavirus
Keywords: COVID-19; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — itolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be blinded to all study staff that has direct access to the subjects and the sponsor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EQ001 (Experimental): EQ001 administered in a blinded fashion by intravenous infusion on Day 1 and Day 8 for a total of 2 doses.
  Interventions: Biological: EQ001
- EQ001 Placebo (Placebo Comparator): Placebo administered in a blinded fashion by intravenous infusion on Day 1 and Day 8 for a total of 2 doses.
  Interventions: Biological: EQ001 Placebo

INTERVENTIONS:
Biological: EQ001 — itolizumab [Bmab600]
  Other Names: itolizumab; Bmab600
  Arms: EQ001
Biological: EQ001 Placebo — EQ001 Placebo
  Arms: EQ001 Placebo

SUMMARY:
This is a randomized controlled trial to evaluate the efficacy and safety of itolizumab in subjects hospitalized with COVID-19.

DETAILED DESCRIPTION:
This study will randomize up to 800 subjects in a 1:1 ratio; itolizumab vs. placebo. Subjects will receive either itolizumab or placebo administered intravenously on Day 1 and Day 8 with follow-up to Day 90. Two interim analyses of futility are planned. The first will take place when approximately 20% of the subjects have been evaluated for the primary endpoint, and the second will take place when approximately 50% of the subjects have been evaluated for the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing and able to, or has a legally acceptable representative who is willing and able to, provide informed consent to participate and to cooperate with all aspects of the protocol.
2. Is male or female, age ≥18 years
3. Is hospitalized with COVID-19 pneumonia with a diagnosis of SARS-CoV-2 infection confirmed by reverse transcriptase polymerase chain reaction (RT-PCR) or equivalent local test within 14 days of randomization.
4. Has PaO2/FiO2 ratio of ≤200 (or equivalent SpO2/FiO2 ratio ~235 within 24 hours before randomization. This ratio may be adjusted based on altitude.

Exclusion Criteria:

1. Has known severe allergic reactions to mAbs.
2. Has active TB or known history of inadequately treated latent or active TB.
3. Has any known active systemic or pulmonary bacterial, fungal, or viral (other than SARS-CoV-2) infection at the time of randomization.
4. Has known active, uncontrolled hepatitis B or hepatitis C or severe liver function impairment from any etiology, as defined by Child-Pugh Class C.
5. Has human immunodeficiency virus (HIV) with known CD4 counts <0.2 × 10^9/L.
6. Has a history of clinically significant cardiac abnormality within 6 months prior to randomization, such as myocardial infarction or stroke, New York Heart Association class III or IV, or clinically significant abnormalities of electrocardiogram (ECG) or cardiac function.
7. Has been on mechanical ventilation for longer than 48 hours during their first continuous episode since admission, is on their second or greater episode of mechanical ventilation at the time of randomization during the concurrent hospitalization, or has received extracorporeal membrane oxygenation (ECMO).
8. Has a declining clinical status with an expected survival <3 days in the opinion of the Investigator.
9. Has received any systemic immunomodulatory or immunosuppressant agents for any condition within 3 months prior to randomization. (Note: a stable, oral, low dose of corticosteroids [prednisone or equivalent ≤10 mg/day] for a chronic condition or any dose of systemic corticosteroids for current COVID-19 treatment are permitted. Local/topical treatments are also permitted.)
10. Has received any biologic treatment for any acute (eg, COVID-19) or chronic conditions (eg, TNFα inhibitors, anti-IL17A, tocilizumab, anti-cytokines, etc.) within 3 months prior to randomization.
11. Is participating in another clinical study of an investigational product and/or received an investigational product within 30 days or within 5 half-lives (whichever is longer) prior to randomization.
12. Is pregnant or breastfeeding, or has a positive pregnancy serum or urine test during Screening.
13. Does not agree to use contraception in the event of sexual activity for 130 days (+90 days for male subjects) after the last dose of study drug if a female of childbearing potential or a male with a partner of childbearing potential. Note: this criterion does not apply to subjects in same-sex relationships.
14. Has inadequate hematologic function during Screening defined as follows:

    * Absolute neutrophil count (ANC) <1.0 × 109/L.
    * ALC <0.5 × 109/L.
15. Requires renal dialysis, either acute or chronic, at the time of randomization.
16. Has a medical, psychiatric, or other condition or circumstance that, in the opinion of the Investigator, could affect the subject's safety, the subject's participation in the study, or the reliability of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who have recovered at Day 28. | Day 28
  Proportion of subjects who have recovered at Day 28.

SECONDARY OUTCOMES:
Proportion of subjects deceased or requiring mechanical ventilation at Day 28. | Day 28
  Proportion of subjects deceased or requiring mechanical ventilation at Day 28.
Proportion of subjects deceased at Day 28. | Day 28
  Proportion of subjects deceased at Day 28.

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs). | Day 90
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE)
Time to maximum itolizumab serum concentration, Tmax | Day 28
  Time to maximum itolizumab serum concentration, Tmax
Maximum itolizumab serum drug concentration, Cmax | Day 28
  Maximum itolizumab serum drug concentration, Cmax
Total itolizumab exposure across time, AUC (from zero to last) | Day 28
  Total itolizumab exposure across time, AUC (from zero to last)
Inflammatory biomarkers | Day 28
  Including but not limited to IL-1, IL-6, IL-17, TNF-α.
Pharmacodynamic markers | Day 28
  sCD6, sALCAM

CONTACTS AND LOCATIONS:
Overall Officials: Maple Fung, MD, Study Director — Equillium
Locations (1):
- Inv Site CO01, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company website — https://equilliumbio.com/